CLINICAL TRIAL: NCT06238050
Title: NOrmoBaric Oxygen Therapy Use In Critical Limb ISchemia
Acronym: NOBILIS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC22_0236; 2023-A02581-44 (Other: ANSM)
Record Dates: First submitted 2022-11-28; First posted 2024-02-02 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Critical Ischemia Limb
Keywords: oxygen therapy
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hospitalized patients suspected of chronic permanent ischemia realizing transcutaneous oxymetry: hospitalized patients suspected of chronic permanent ischemia realizing transcutaneous oxymetry are enroled in the study.
  The WIfI score is calculated at the inclusion.
  Interventions: Procedure: introduction of oxygen therapy or not

INTERVENTIONS:
Procedure: introduction of oxygen therapy or not — During hospitalisation, surgeon decides if patient needs and will have an oxygen therapy during this hospitalisation and at home.

SUMMARY:
Peripheral arteriopathy disease (PAD) affects 1 million people in France. In its most advanced stage: chronic permanent ischemia also called critical ischemia, the prognosis of patients is burdened with a one-year mortality rate of 30%. Chronic permanent ischemia results from a lack of oxygen supply to the microcirculatory network, responsible for tissue death and the development of trophic disorders. In this context, many studies have focused on the contribution of hyperbaric oxygen therapy, however none demonstrates with certainty its beneficial effect with a heavy set-up for teams and patients. Furthermore, it appears that normobaric oxygen therapy could have its place in this context by temporarily restoring a sufficient level of transcutaneous oxygen. However, even if normobaric oxygen therapy is common practice although empirical for some practitioners, no data demonstrates its real interest. The purpose of this study is therefore to report the proportion, in usual practice, of patients with permanent chronic ischemia of the lower limb(s), benefiting from normobaric oxygen therapy, but also to show the interest of the contribution of this therapy in usual comprehensive management of these patients. This is a pilot study, after which, if the hypothesis is confirmed, it may be proposed to carry out a randomized study, on a large scale, in order to validate the use of normobaric oxygen therapy in the context of chronic permanent ischemia.

DETAILED DESCRIPTION:
In arterial pathology of the lower limbs at the stage of chronic permanent ischemia, very few data exist on the benefit of normobaric oxygen therapy in these patients. The purpose of the present study is to report the proportion in usual practice of patients benefiting from normobaric oxygen therapy and to show the interest of the contribution of this therapy in the usual global management of patients presenting with chronic permanent ischemia of the lower limbs.

Regarding the Wound, Ischemia, Foot Infection Score (WIfI score), it includes three sub-parts, each of which has a specific evaluation grid scoring between 0 and 3. From this evaluation grid, an overall score can be calculated with different interpretations to determine the risk of amputation at one year as well as the probability of improvement in the event of revascularization, ranging from very low risk to high risk. Nevertheless, the overall evaluation of the score could mask a significant improvement in one of the items evaluated, impacting the clinical management and the future of the patient. This is why, during this study, the improvement of each item of the WIfI score separately will be studied.

The hypothesis is that putting patients in chronic permanent ischemia on oxygen therapy, which is performed frequently, brings a medical benefit compared to patients who do not benefit from it.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in the recruiting centre.
* Patient fulfilling the clinical and paraclinical criteria (resting TcpO2 values < 30mmHg) of the definition of chronic permanent ischemia with or without trophic disorders.

Exclusion Criteria:

* Patient suffering from acute or decompensated heart or respiratory failure.
* Patient suffering from chronic obstructive pulmonary disease (COPD) stage III or IV.
* Patient with allergies to medical adhesives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized patient with symptoms of chronic permanent ischemia
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of clinical characteristics of patients, whether or not they benefit from oxygen therapy in usual practices. | 6 months
  Determination of patients' characteristic with or without a prescription of oxygen therapy to inventorized clinical practices.
Comparison of biological characteristics of patients, whether or not they benefit from oxygen therapy in usual practices. | 6 months
  Determination of patients' characteristics with or without a prescription of oxygen therapy to inventorized clinical practices.

SECONDARY OUTCOMES:
Collection of all investigations carried out since inclusion and all modifications of medical therapy or implementation of surgical treatment. | 6 months
  Descriptive study of investigations and therapies (medical and surgical) carried out during the patient's follow-up period
prevalence of decision-making parameters by using the sheet sent to the prescribing doctor by the patient. | 6 months
  Descriptive study of the parameter(s) which allowed the prescriber to make the decision to implement oxygen therapy.
difference in the WIfI score items at inclusion and at 6 months. | 6 months
  Evaluation of the evolution of chronic permanent ischemia according to the administration in current practice of normobaric oxygen therapy.
All-cause mortality at 6 months. | 6 months
  Evaluation of the evolution of chronic permanent ischemia according to the administration in current practice of normobaric oxygen therapy.
occurrence of an amputation between one week after inclusion and 6 months. | 6 months
  Evaluation of the evolution of chronic permanent ischemia according to the administration in current practice of normobaric oxygen therapy.
difference in score obtained at 1 month and at 6 months depending on the presence of chronic permanent ischemia or not and the administration of oxygen or not. | 1 and 6 month
  Assessment of the quality of life of patients suspected of chronic permanent ischemia using the Vascu-QOL-6 questionnaire
Proportion of compliant patients in whom oxygen was prescribed on an outpatient basis | 1 and 6 month
  Evaluation of compliance with oxygen for patients benefiting from it

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - University Hospital, Angers
  - Hospital Center, Cholet
  - Hospital Center, Le Mans